CLINICAL TRIAL: NCT05558085
Title: A Cost-Benefit Analysis of EFNEP Utilizing Biomarkers of Chronic Disease Risk
Brief Title: Biomarker Cost-Benefit Analysis of EFNEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Dakota State University (Other)
Collaborators: University of Idaho (Other); University of Maryland, College Park (Other); Washington State University (Other); Michigan State University (Other); Colorado State University (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1843412-1
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Disease
Keywords: Diet; Nutrition Education; Biomarker; Cost-benefit analysis; EFNEP
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFNEP Group (Experimental): Subjects will receive the EFNEP Eat Smart Being Active class series.
  Interventions: Behavioral: Expanded Food and Nutrition Education Program (EFNEP)
- Control Group (No Intervention): Subjects will receive no EFNEP intervention.

INTERVENTIONS:
Behavioral: Expanded Food and Nutrition Education Program (EFNEP) — Subjects will participate in nine hands-on EFNEP lessons to teach nutrition, healthy lifestyle choices, physical activity, food preparation, food safety, and food resource management.
  Arms: EFNEP Group

SUMMARY:
The goal of this integrated project is to assess whether EFNEP is a cost-effective nutrition education intervention that generates sustained improvement in chronic disease biomarkers. This project will be unique in its use of objective biomarkers, instead of self-reported behaviors, to quantify the economic benefits generated by EFNEP through chronic disease prevention. A paired location untreated control group quasi-experimental design will be employed, with biomarkers (BMI, blood pressure, HbA1c) measured for 500 adults across four representative state EFNEP programs (CO, FL, MD, WA). Biomarkers will be measured pre-EFNEP, 6-months-post-EFNEP and 1-year-post-EFNEP. Analytical techniques will include cost-benefit, bivariate, and multivariate analyses.

DETAILED DESCRIPTION:
According to the CDC, 60% of US adults have a diagnosed chronic disease. This indicates the need for focused efforts to change modifiable risk factors including diet and exercise. The Expanded Food and Nutrition Education Program (EFNEP) aims to prevent chronic diseases by educating and encouraging vulnerable populations to adopt a healthy diet and physical activity. Addressing the program priority area Diet, Nutrition and the Prevention of Chronic Diseases, the long-term goal of this integrated project is to assess whether EFNEP is a cost-effective nutrition education intervention that generates sustained improvement in chronic disease biomarkers. This project will be unique in its use of objective biomarkers, instead of self-reported behaviors, to quantify the economic benefits generated by EFNEP through chronic disease prevention.

Project research objectives include analyzing EFNEP's sustained impact on chronic disease biomarkers and developing and applying a biomarker-based cost-benefit analysis methodology. Extension objectives are to develop an online cost-benefit analysis tool and webinar for nutrition education program evaluation. Education objectives are to provide graduate students with experiential learning opportunities in data collection and analysis.

A paired location untreated control group quasi-experimental design will be employed, with biomarkers (BMI, blood pressure, HbA1c) measured for 500 adults across four representative state EFNEP programs (CO, FL, MD, WA). Biomarkers will be measured pre-EFNEP, 6-months-post-EFNEP and 1-year-post-EFNEP. Analytical techniques will include cost-benefit, bivariate, and multivariate analyses. Project results will expand the EFNEP knowledge-base, allowing for program content and delivery modifications that maximize the impact of taxpayer dollars allocated to chronic disease prevention.

ELIGIBILITY:
Inclusion Criteria:

* Free-Living
* Speaks and understands English and/or Spanish
* Income at or below 185% of the Federal Poverty Line

Exclusion Criteria:

* Being pregnant, nursing, and/or less than 9-months postpartum

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Height from Baseline to 6 Months Post Intervention | Change in height measurement from baseline to 6 months post intervention
  Height (m) is measured using a portable stadiometer.
Change in Height from Baseline to 12 Months Post Intervention | Change in height measurement from baseline to 12 months post intervention
  Height (m) is measured using a portable stadiometer.
Change in Weight from Baseline to 6 Months Post Intervention | Change in weight measurement from baseline to 6 months post intervention
  Weight (kg) is measured using a portable scale.
Change in Weight from Baseline to 12 Months Post Intervention | Change in weight measurement from baseline to 12 months post intervention
  Weight (kg) is measured using a portable scale.
Change in Systolic and Diastolic Blood Pressure from Baseline to 6 Months Post Intervention | Change in Systolic and Diastolic blood pressure measurements from baseline to 6 months post intervention
  Systolic and Diastolic blood pressure are measured using an OMRON Silver blood pressure monitor
Change in Systolic and Diastolic Blood Pressure from Baseline to 12 Months Post Intervention | Change in Systolic and Diastolic blood pressure measurements from baseline to 12 months post intervention
  Systolic and Diastolic blood pressure are measured using an OMRON Silver blood pressure monitor
Change in HbA1c from Baseline to 6 Months Post Intervention | Change in HbA1c measurement from baseline to 6 months post intervention
  HbA1c is measured using A1CNow monitor.
Change in HbA1c from Baseline to 12 Months Post Intervention | Change in HbA1c measurement from baseline to 12 months post intervention
  HbA1c is measured using A1CNow monitor.

SECONDARY OUTCOMES:
Change in EFNEP Adult Questionnaire Responses Baseline to 6 Months Post Intervention | Change in EFNEP Adult Questionnaire Responses Baseline to 6 Months Post Intervention
  The EFNEP Adult Questionnaire includes questions regarding food and physical activity behaviors.
Change in EFNEP Adult Questionnaire Responses Baseline to 12 Months Post Intervention | Change in EFNEP Adult Questionnaire Responses Baseline to 12 Months Post Intervention
  The EFNEP Adult Questionnaire includes questions regarding food and physical activity behaviors.
Change in 24-Hour Dietary Recalls Baseline to 6 Months Post Intervention | Change in 24-Hour Dietary Recalls Baseline to 6 Months Post Intervention
  24-hour dietary recalls will be administered to capture change in food and beverage intake.
Change in 24-Hour Dietary Recalls Baseline to 12 Months Post Intervention | Change in 24-Hour Dietary Recalls Baseline to 12 Months Post Intervention
  24-hour dietary recalls will be administered to capture change in food and beverage intake.
Participant Demographics Baseline | Baseline.
  A range of participant demographics will be collected including sex, age, race/ethnicity, public assistance receipt, pregnancy status, and breastfeeding status.
Participant Demographics Post Intervention | Immediately Post Intervention.
  A range of participant demographics will be collected including public assistance receipt, pregnancy status, and breastfeeding status.
Participant Demographics 6 Months Post Intervention | 6 Months Post Intervention
  A range of participant demographics will be collected including public assistance receipt, pregnancy status, and breastfeeding status.
Participant Demographics 12 Months Post Intervention | 12 Months Post Intervention
  A range of participant demographics will be collected including public assistance receipt, pregnancy status, and breastfeeding status.
Participant Health Status Baseline | Baseline
  A Health Questionnaire will be used to identify whether participants have a health condition, take medication(s) for a health condition, and smoke.
Participant Health Status 6 Months Post Intervention | 6 Months Post Intervention
  A Health Questionnaire will be used to identify whether participants have a health condition, take medication(s) for a health condition, and smoke.
Participant Health Status 12 Months Post Intervention | 12 Months Post Intervention
  A Health Questionnaire will be used to identify whether participants have a health condition, take medication(s) for a health condition, and smoke.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Colorado State University, Fort Collins, Colorado
  - University of Florida, Gainesville, Florida
  - University of Maryland, College Park, Maryland
  - Washington State University, Pullman, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available on South Dakota State University's Open Access Institutional Repository, Open PRAIRIE.